CLINICAL TRIAL: NCT07353021
Title: Clinical Trial on Long-Term Effects of a Biofield Patch on Anxiety, Sleep, and Energy. A Randomized Double-Blind Placebo-Controlled 4-week Trial.
Brief Title: Longterm Effects of a Biofield Patch on Anxiety, Sleep, and Energy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 206-008
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Sleep
Keywords: Sleep; Stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled study design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will use an active biofield patch daily for 4 weeks. The active biofield patch will look identical to a placebo patch, and will be blinded.
  Interventions: Device: Active dermal patch
- Group 2 (Experimental): Participants will use a placebo patch daily for 4 weeks. The placebo patch will look identical to an active patch, and will be blinded.
  Interventions: Device: Placebo patch

INTERVENTIONS:
Device: Active dermal patch — Non-transdermal patch
  Arms: Group 1
Device: Placebo patch — Non-transdermal patch
  Arms: Group 2

SUMMARY:
The goal for this clinical trial is to compare an active biofield non-transdermal skin patch to a placebo patch in people who frequently experience anxiety.

DETAILED DESCRIPTION:
The goal for this clinical trial is to document effects of a photobiomodulating non-transdermal patch compared to a placebo patch, in a randomized double-blind placebo-controlled design.

Data on stress and anxiety levels will be collected using the GAD and OASIS questionnaires as well as the Warwick-Edinburgh Mental Wellbeing Scales collected. The data collected will show whether the daily use of the patch leads to a change in general self-reported stress and anxiety levels. Data on energy levels will be collected using a Wellness questionnaire. Data on sleep quality will be collected using the Leeds sleep evaluation questionnaire, to document whether using the active patch impacts self-reported sleep.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of all genders;
* Age 18-75 years (inclusive);
* BMI between 18.0 and 34.9 (inclusive)
* Experiencing intermittent episodes of anxiety on a regular basis, leading to either avoiding specific situations, or experiencing stress both in anticipation of, and during such situations.

  * Specific situations that occur regularly that cause anxiety, for example:

    * Performing specific tasks at work or at home;
    * Inter-personal conflicts at work or at home;
    * Driving or commuting;
    * Fearful and worrying about one's own situation (such as paying bills);
    * Worrying about ongoing problems experienced by others.

Exclusion Criteria:

* Cancer during past 12 months;
* Chemotherapy during past 12 months;
* Currently taking anxiolytic, hypnotic, or anti-depressant prescription medication;
* Currently taking nutritional supplements judged by the study coordinator to negate or camouflage the effects of the test product;
* Participation in another clinical trial study during this trial, involving an investigational product or lifestyle change;
* Serious active illness within past 6 months;
* People who are pregnant, nursing, or trying to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
General Anxiety Disorder 7 (GAD 7) Questionnaire | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Change from baseline in anxiety score using the General Anxiety Disorder 7-item. The General Anxiety Disorder-7 scale evaluates anxiety severity using scores ranging from 0-21, where higher scores indicate higher anxiety severity.

SECONDARY OUTCOMES:
Overal Anxiety Severity and Impairment Scale (OASIS) Questionnaire | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Change from baseline in Overall Anxiety Severity and Impairment Scale (OASIS) score. The Overall Anxiety Severity and Impairment scale evaluates anxiety and impact on daily living in participants with a score between 0 and 25, where higher scores indicate higher anxiety severity and impact on daily living.

OTHER OUTCOMES:
Warwick-Edinburgh Mental Wellbeing Scale | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Changes from baseline in mental wellbeing using the Warwick-Edinburgh Mental Wellbeing scale. The Warwick-Edinburgh Mental Wellbeing scale evaluates self reported happiness and satisfaction as well as psychological functioning, good relationships with others, and self realization.
Wellness Questionnaire | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Change from baseline in wellness evaluated using a Wellness questionnaire. The Wellness questionnaire consists of 30 questions, generating scores for physical, mental functioning, emotional wellbeing, stress, social functioning, sleep, and energy/vitality, where higher scores reflect better wellness.
Leeds Sleep Questionnaire | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks.
  Changes from baseline in sleep quality. The Leeds Sleep Evaluation Questionnaire is a 10 item linear-log scale based on questions across several domains of sleep, where higher scores reflect better sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States